CLINICAL TRIAL: NCT04930185
Title: Reducing Vaccine Hesitancy (VH) And Vaccine Refusal (VR): Its' Correlation Factors and an Educational Intervention Programme
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunway University (Other)
Responsible Party: Principal Investigator, Ooi Pei Boon, Principal Teaching Fellow, Sunway University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SRB/IIR/SMC/F/21/001
Record Dates: First submitted 2021-06-03; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: COVID-19 Vaccination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pamphlet (Experimental): Participants will received pamphlet about COVID-19 vaccination
  Interventions: Behavioral: Reducing Vaccine Hesitancy (VH) And Vaccine Refusal (VR): An Educational Intervention Programme
- Webinar (Experimental): Participants will received webinar about COVID-19 vaccination
  Interventions: Behavioral: Reducing Vaccine Hesitancy (VH) And Vaccine Refusal (VR): An Educational Intervention Programme
- SMS (Experimental): Participants will received SMS about COVID-19 vaccination
  Interventions: Behavioral: Reducing Vaccine Hesitancy (VH) And Vaccine Refusal (VR): An Educational Intervention Programme

INTERVENTIONS:
Behavioral: Reducing Vaccine Hesitancy (VH) And Vaccine Refusal (VR): An Educational Intervention Programme — Participants will be receiving the pamphlet about the COVID-19 vaccination information during the intervention.
  They will received 3 different sets of questionnaire to measured their level of vaccine hesitancy and vaccine refusal in 3 different time points: (a) before intervention, (b) after the intervention, and (c) 3 months after the intervention.
  Data cleansing will be conducted based on the per-protocol analysis. Pre-protocol is a comparison of treatment groups that includes only those patients who completed the treatment originally allocated.
  Arms: Pamphlet
Behavioral: Reducing Vaccine Hesitancy (VH) And Vaccine Refusal (VR): An Educational Intervention Programme — Participants will be receiving the webinar last for half an hour about the COVID-19 vaccination information during the intervention.
  They will received 3 different sets of questionnaire to measured their level of vaccine hesitancy and vaccine refusal in 3 different time points: (a) before intervention, (b) after the intervention, and (c) 3 months after the intervention.
  Data cleansing will be conducted based on the per-protocol analysis. Pre-protocol is a comparison of treatment groups that includes only those patients who completed the treatment originally allocated.
  Arms: Webinar
Behavioral: Reducing Vaccine Hesitancy (VH) And Vaccine Refusal (VR): An Educational Intervention Programme — Participants will be receiving the SMS about the COVID-19 vaccination information during the intervention.
  They will received 3 different sets of questionnaire to measured their level of vaccine hesitancy and vaccine refusal in 3 different time points: (a) before intervention, (b) after the intervention, and (c) 3 months after the intervention.
  Data cleansing will be conducted based on the per-protocol analysis. Pre-protocol is a comparison of treatment groups that includes only those patients who completed the treatment originally allocated.
  Arms: SMS

SUMMARY:
The COVID-19 pandemic has spread to over 200 countries worldwide and is still on the rise in 88 countries. Unfortunately, Malaysia is not the exception and registered 340,642 COVID-19 cases till 29 March 2021 since the outbreak of the pandemic.

COVID-19 virus can be transmitted from an infected person to others through droplets when coughing or sneezing as well as by touching objects infected with the virus. Although precautionary measures, which include the regular and mandatory use of face masks, reducing crowds, and physical distancing, have been widely encouraged by WHO and the Malaysian government, getting COVID-19 vaccination remain the way forward to curb the wide spread of the virus and to return to the normal.

However, the public awareness on the importance of getting vaccinated is still low with high level of vaccination hesitance and refusal. In Malaysia, this challenge is compounded further due to a lack of COVID-19 vaccination educational intervention programme in Bahasa Malaysia to educate the predominantly larger group in the population who are more conversant in ther national language. In order to improve the acceptance rate towards the COVID-19 vaccination in Malaysia, it is imperative to design a comprehensive intervention program that will increase the awareness and knowledge with regards to the efficacy of the COVID-19 vaccine as a solution in overcoming this pandemic.

With this in mind, this study aims to identify the correlational factors of COVID-19 and develop an educational intervention programme on COVID-19 vaccination and thereafter, assess the effectiveness of this educational intervention programme.

DETAILED DESCRIPTION:
Research Objectives

1. Examine the association among vaccination intention, attitudinal belief, subjective norms, perceived behavioral control, vaccine hesitancy and its reasons among the Malaysian population.
2. Develop an educational intervention Programme on COVID-19 vaccination to increase knowledge, positive attitudes, and acceptance toward COVID-19 vaccination
3. Assess the effectiveness of the educational intervention programme

Research Hypothesis

The hypotheses are:

1. The Ministry of Sciences and Technology (2021) reported that the percentage of Malaysians who voluntarily registered for the COVID-19 vaccine is still low. The researcher, therefore, hypothesize that the level of knowledge, positive attitudes, and acceptance towards the COVID-19 vaccine among Malaysian population to be rather low.
2. The researcher hypothesize that there is an association among vaccination intention, attitudinal belief, subjective norms, perceived behavioral control, vaccine hesitancy and its reasons among the Malaysian population
3. The researcher hypothesize that the educational intervention programme has a statistically significant effect on reducing vaccination hesitancy and vaccination refusal between the baseline and the assessment soon after the program as well as at 3 months after the programme as compared to the control group)

The Study There are 2 phases in this study. Phase 1 is the cross-sectional study, while Phase 2 will look into the programme development and feasibility and the implementation of a cluster randomised controlled trial (RCT).

Phase 1 Cross-sectional Study

Study design & procedure:

1. This cross-sectional study will utilize both online and paper questionnaire.
2. The sample will be recruited through both voluntary response sampling and snowball sampling methods. The survey will be sent out to Malaysian who are more than 18 years old in the online social media platforms.
3. To ensure the cross-sectional study to be effective, the researcher decided our sample size based on Krejcie & Morgan (1970) method that has commonly and widely been used in simple random sampling studies for each sample. Thus, for a wide of 32 million of population in Malaysia, the researcher had targeted for a total of 384 participants are sufficient.
4. This cross-sectional study aims to examine the association among vaccination intention, attitudinal belief, subjective norms, perceived behavioural control, vaccine hesitancy and its reasons among the Malaysian population.

Study site and participants

1. The cross-sectional study will be taking place in online setting. A few social media platforms are chosen for this purpose such as Facebook, Instagram, WhatsApp, and et-cetera.
2. Recruitment materials and survey will be shared on the social medial platforms and advocate public to share among others who are eligible.

Phase 2 (a): Programme Development and Feasibility Study

Study design & procedure:

1. A group of experts consisting of public health experts in health education, health psychology, and other health-care providers (communicable disease background) will hold online meetings (Focus Group Discussions) to develop the modules for the Programme based on literature review, best practices in the field and in consultation with public health experts and other ministerial departments.
2. For a focus group discussion (FGD) to be effective, the number of participants shall between 6-8 per group (Krueger & Casey, 2002). The researcher will target 8 per group and organize up to 5 groups and/or when the researcher reach data saturation points.
3. The FGDs will aim to build the content and activities of the Programme. The core members of this research team will finalise the Programme structure, before holding a second online meeting with the experts involved to confirm its validity. This Programme will continue to be refined throughout the study based on the feasibility study results.

Phase 2 (b): Cluster Randomised Controlled Trial (RCT).

Study design & procedure:

1. To evaluate the effectiveness of the Programme, a cluster randomised controlled trial with three assessment points (Baseline, immediate after intervention and 3-month follow-up) will be conducted with the materials and outcome measures listed.
2. This will be a study based on pre/post multiple time series study design.
3. Students from the School of Medical & Life Sciences, Sunway University, Faculty of Social Sciences, Quest University International, Ipoh and Centre of Community Health Studies, UKM will be engaged in the design and development of the approved content. By doing so, students from various universities would have a chance to apply what they have learned in the classrooms into the real life.
4. Materials will be in the form of pamphlet, webinar content and SMS and in Bahasa Malaysia.

Sample size calculation:

1. Non-inferiority designed will be used to show that the new treatment is as effective but need not superior when compared to the standard treatment (Zhong, 2009).
2. For non-inferiority design, the formula is:
3. Based on the recent published results, non-response rate of standard vaccine rate is reported to be 7% (Khubchandani et al., 2021). Thus, sample size required would be:

   * N= 2 x [(1.645+0.845)/0.1]2 x 0.07 x (1-0.07)
   * N= 80.7 (approximately 81 participants)
4. Assuming a dropout rate of 20%, the researcher will recruit at least 100 participants in each category for each education material used, making a total of 300 for each site (Figure 1).

Study site and participants

1. The cluster randomised controlled trial with three parallel arms (i.e., 3 intervention groups ) will be performed in both West and East Coast Malaysia. One major health facility/university will be selected and approached.
2. Recruitment materials designed will be shared and distributed both online and offline to the health facilities, schools, churches, mosques, temples, NGOs, recreation malls and societies.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years and above
* Able to provide informed consent (verbal/written) to participate
* Understand either Bahasa Malaysia
* Participants who have not received their COVID-19 vaccination
* Participants who have access to smart phone and/or mobile phone
* Participants who have access to internet.

Exclusion Criteria:

* Those who have had any prior history of psychological or neurological illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Reducing Vaccine Hesitancy | 17 months
  The vaccine hesitancy scale

SECONDARY OUTCOMES:
Reducing Vaccine Hesitancy | 17 months
  The researcher will build a dichotomous scale from ground up to see the acceptance rate of participants towards each brand of vaccine available in Malaysia

CONTACTS AND LOCATIONS:
Locations (1):
- Sunway University, Petaling Jaya, Selangor, Malaysia